CLINICAL TRIAL: NCT06879938
Title: Concomitant Treatment with Topical Hyaluronic Acid and High Concentration Oxygen Therapy (Vaginal Natural Oxygenation Device - VNOD) in the Improvement of Symptoms Related to Genitourinary Syndrome of Menopause in Women with Natural and Oncological Postmenopause: Open-Label, Single-Center, Randomized Study
Brief Title: Concomitant Treatment with Topical Hyaluronic Acid and High Concentration Oxygen Therapy (Vaginal Natural Oxygenation Device - VNOD) in the Improvement of Symptoms Related to Genitourinary Syndrome of Menopause in Women with Natural and Oncological Postmenopause: Open-Label, Single-Center, Randomize
Acronym: Caress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Rossella Nappi, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Caress
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Genitourinary Syndrome of Menopause

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-concentration vaginal oxygen therapy (Caress Flow) with topical hyaluronic acid (Experimental)
  Interventions: Device: High-concentration vaginal oxygen therapy (Caress Flow) with topical hyaluronic acid
- Hyaluronic acid-based gel (Hydeal-D®) applied once every three days (Active Comparator)
  Interventions: Device: hyaluronic acid-based gel (Hydeal-D®)

INTERVENTIONS:
Device: High-concentration vaginal oxygen therapy (Caress Flow) with topical hyaluronic acid — five treatment sessions of high-concentration vaginal oxygen therapy (Caress Flow) with topical hyaluronic acid 2 weeks apart with a duration of approximately 15 minutes
  Arms: High-concentration vaginal oxygen therapy (Caress Flow) with topical hyaluronic acid
Device: hyaluronic acid-based gel (Hydeal-D®) — hyaluronic acid-based gel (Hydeal-D®) applied once every three days for 12 weeks
  Arms: Hyaluronic acid-based gel (Hydeal-D®) applied once every three days

SUMMARY:
The Caress study is a single-center, open-label, randomized controlled trial (RCT) evaluating the efficacy of a combined treatment using topical hyaluronic acid and high-concentration oxygen therapy (Vaginal Natural Oxygenation Device - VNOD) in improving symptoms of Genitourinary Syndrome of Menopause (GSM) in postmenopausal women, including those with a history of breast cancer. The primary objective is to assess vaginal dryness improvement one month after treatment, comparing two groups: an experimental group receiving VNOD therapy with hyaluronic acid and a control group using a hyaluronic acid-based gel (Hydeal-D®). Secondary endpoints include the evaluation of additional vaginal symptoms (pain, irritation, itching, sexual health, quality of life) up to six months post-treatment. The study will enroll 80 women (40 with a history of breast cancer and 40 without). Statistical analysis will use chi-square tests and logistic regression to compare symptom severity reduction between the two groups. With a duration of 18 months, the study aims to provide an innovative, non-hormonal treatment option to improve the quality of life for postmenopausal women, particularly those with a history of breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signature
* Willingness to undergo treatment and follow-up evaluations according to the schedule outlined in the protocol
* Age > 18 years

Cohort 1:

* Diagnosis of non-metastatic breast cancer (M0/Mx according to TNM system) who have undergone surgical and/or chemotherapy and/or immunotherapy and/or radiotherapy and/or endocrine treatment.
* Postmenopausal women (FSH > 30 UIIU/L, E2 < 20 pg/ml), either naturally or surgically induced, or iatrogenic post-chemotherapy with absent menstrual cycle for at least 6 months; or premenopausal women on treatment with LHRH analog +/- tamoxifen and/or aromatase inhibitor for at least 6 months.
* At least a score of 2 (moderate) for vaginal dryness associated with vulvovaginal atrophy (score 2-3 on the MBS scale).
* Signs of pelvic static alterations not exceeding POP-Q score 2 (POP-Q).

Cohort 2:

* Postmenopausal women (FSH > 30 UI/L, E2 < 20 pg/ml), with absent menstrual cycle for at least 6 months, or women who have undergone bilateral adnexectomy at least 6 months ago.
* At least a score of 2 (moderate) for vaginal dryness associated with vulvovaginal atrophy (score 2-3 on the MBS scale).
* Signs of pelvic static alterations not exceeding POP-Q score 2 (POP-Q).

Exclusion Criteria:

* Other current therapy aimed at resolving symptoms associated with vulvo-vaginal atrophy, with the exception of the use of lubricants if sexual activity is present;
* HRT in progress or discontinued for less than 6 months;
* Ongoing vulvo-vaginal and urinary infections;
* Bleeding of ndd;
* Pathological pap-test within the previous 12 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
vaginal dryness one month after the completion of treatment | one month
  comparison of the two treatment arms for the percentage of patients with a moderate or severe degree of vaginal dryness according to the Most Bothersome Symptoms - MBS scale (scores 2-3) one month after the end of treatment in the total enrolled women (Cohort 1 + Cohort 2).

SECONDARY OUTCOMES:
treatment compliance | one month
  Comparison of the percentage of patients who, at the visit conducted one month after the completion of treatment, report not having followed the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SSD Ostetricia e Ginecologia 2 - Riproduzione e Procreazione Medicalmente Assistita, Pavia, Pavia, Italy